CLINICAL TRIAL: NCT06569173
Title: Comparison of the Drainage/Anti-reflux Effect and Stent-Related Symptoms Between Anti-Reflux Stents and Standard DJ Stents in Children With Urolithiasis
Brief Title: Comparison of Stent-Related Symptoms Between Anti-Reflux Stents and Standard DJ Stents in Children With Urolithiasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Hongbo Liu, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-IRB-0212-IR-01
Record Dates: First submitted 2024-07-23; First posted 2024-08-23 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Urolithiasis; Child, Only
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LaiKai Anti-Reflux Ureteral Stent (19903) (Experimental): LaiKai Anti-Reflux Ureteral Stent (19903) arm received anti-reflux stent.
  Interventions: Device: LaiKai anti-reflux ureteral stent
- LaiKai Ureteral Stent (92001024) (Active Comparator): LaiKai Ureteral Stent (92001024) arm received regular ureteral stent.
  Interventions: Device: LaiKai Ureteral Stent

INTERVENTIONS:
Device: LaiKai anti-reflux ureteral stent — Ureteral stents are serving to support the ureter and facilitate urine drainage with an anti-reflux valve.
  Arms: LaiKai Anti-Reflux Ureteral Stent (19903)
Device: LaiKai Ureteral Stent — Ureteral stents are serving to support the ureter and facilitate urine drainage.
  Arms: LaiKai Ureteral Stent (92001024)

SUMMARY:
The aim of this study is to investigate the effectiveness and related complications of anti-reflux stents used in pediatric urolithiasis surgery at the Children's Hospital affiliated with Zhejiang University School of Medicine, by comparing them with conventional stents.

DETAILED DESCRIPTION:
Ureteral stents are crucial adjunctive devices following urolithiasis surgery, serving to support the ureter and facilitate urine drainage. However, the application of these stents can lead to complications such as urinary tract infections, lumbar pain, and bladder irritative symptoms, which significantly impact the quality of life in pediatric patients. Novel designs, such as anti-reflux stents equipped with valves, have been optimized to enhance unidirectional urine flow while effectively preventing retrograde urine flow. It is anticipated that these designs could alleviate symptoms of lumbar pain and urinary tract infections, thereby improving the postoperative recovery quality in children. Current adult studies suggest that anti-reflux stents might reduce urine reflux but may also be associated with significantly stronger urinary symptoms. To date, there have been no pediatric studies reported on the efficacy of anti-reflux stents. The aim of this study is to investigate the effectiveness and related complications of anti-reflux stents used in pediatric urolithiasis surgery at the Children's Hospital affiliated with Zhejiang University School of Medicine, by comparing them with conventional stents.

ELIGIBILITY:
Inclusion Criteria:

1. A definitive diagnosis of urinary tract stones by CT scan, with indications for ureteroscopic lithotripsy (URL), percutaneous nephrolithotomy (PCNL), laparoscopic/open stone extraction with or without robotic assistance, or combined endoscopic lithotripsy, and no contraindications;
2. Age is less than 18 years old;
3. For preschool children, the informed consent form is signed by the parents; for school-age children, the informed consent form is signed by both the parents and the child themselves.

Exclusion Criteria:

1. A history of recurrent bladder irritative symptoms or urinary tract infections;
2. Severe renal insufficiency, anatomical or functional solitary kidney, and other significant comorbidities that render the child unsuitable for participation in the study;
3. Stent placement surgery within the past 3 months;
4. Recent use of medications that may interfere with the study results, such as solifenacin;
5. Stent removal surgery performed at an external medical facility.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-08-23 (Estimated); Study Completion 2025-08-23 (Estimated)

PRIMARY OUTCOMES:
The effect of stents on body pain | Two weeks after stents inserting and two weeks after stents removing
  Inquire whether the child has experienced body pain, especially lumbar pain after the insert or removal of the stent. If yes, assign a value of 1; if no, assign a value of 0. The higher the score, the worse the stent is in terms of relieving lumbar pain.

SECONDARY OUTCOMES:
The effect of stents on stone-free rate | Two weeks after stents inserting and two weeks after stents removing
  Calculate the stone clearance rate for children three months and half a year after surgery. The higher the stone clearance rate, the better the stent's effectiveness.
The effect of stents on urinary symptoms | Two weeks after stents inserting and two weeks after stents removing
  Use a self-administered questionnaire to understand the children's daytime urination intervals, times getting up at night, number of urge urinary incontinence episodes, number of genuine urinary incontinence episodes, times of incomplete urination, times of burning sensation during urination, number of hematuria episodes, degree of hematuria, and overall impact of urinary tract symptoms. Scores are assigned from 1 to 3 or 1 to 5 for different questions, with higher scores indicating poorer stent effectiveness in the corresponding dimension.
The effect of stents on daily activities and psychological well-being | Two weeks after stents inserting and two weeks after stents removing
  Based on the questions in the self-administered questionnaire, including "Does the stent affect daily activities?", "Does the stent affect the child's social interactions?", and "Does the stent cause the child to have feelings of inferiority?", we understand the impact of the stent on the child's daily life and psychological well-being. The results are categorized as "No impact", "Slight impact", and "Significant impact", with corresponding scores of "1-3 points". The higher the score, the greater the adverse effect of the stent on the child.
The effect of stents on clinical presentation | Two weeks after stents inserting and two weeks after stents removing
  Understand the impact of the stent on children's urinary tract infections, antibiotic use, and emergency department visits through a questionnaire. The results are scored as "0-1" or "1-5", with higher scores indicating a greater adverse effect of the stent.
The effect of the stent on learning | Two weeks after stents inserting and two weeks after stents removing
  Understand the impact of the stent on the child's learning situation through a questionnaire, with the results scored on a scale of "0-1". The higher the score, the greater the adverse impact of the stent on learning.

CONTACTS AND LOCATIONS:
Overall Officials: Hongbo Liu, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China